CLINICAL TRIAL: NCT04637867
Title: Multicentre Study on Nosocomial Transmission of SARS-CoV-2 Virus: an Ancillary Study
Brief Title: COVID-19 - Multicentre Study on Nosocomial Transmission of SARS-CoV-2 Virus: an Ancillary Study (NOSO-COR IMMUNO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_0761
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2021-06

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT-PCR confirmed COVID-19 patients (Other): RT-PCR confirmed patients included in the NOSO-COR study are invited six and 12 months after the initial infection to provide blood (41.5mL in total), salivary and nasopharyngeal samples and to complete a questionnaire. Each visit is expected to take about one hour.
  Interventions: Other: Collection of blood, salivary and nasopharyngeal samples.

INTERVENTIONS:
Other: Collection of blood, salivary and nasopharyngeal samples. — Each visit M6 and M12
  * Blood: 1 PAXgene tube (2.5mL) 1 EDTA tube (4mL), 1 dry tube with gel (5mL), 3 EDTA tubes (10mL each)
  * Salivary sample
  * Nasopharyngeal sample

SUMMARY:
There are still uncertainties about the existence of protective immunity and the duration of protective antibodies in patients infected with SARS-CoV-2. Serological testing is an appropriate tool for epidemiological investigations to assess the persistence of antibodies over time. The nature of the immune response induced by this virus is also poorly understood. This ancillary study aims at assessing the immunological characteristics of patients that participated in the NOSO-COR study at Hospices Civils de Lyon six and twelve months after the initial infectious episode.

Two visits will be scheduled at 6 and 12 months (± 1 month) after the initial SARS-CoV-2 infectious episode, Blood, saliva and nasopharyngeal samples will be collected for seroprevalence and immunological investigation.

ELIGIBILITY:
Inclusion Criteria:

SARS-CoV-2 confirmed by RT-PCR

* Adults > 18 years
* Signed consent form
* Affiliated to the French health system

Exclusion Criteria:

* Pregnant women
* Hospitalized patients
* Individuals subject to legal protection
* Imprisoned individuals
* Individuals who have expressed an opposition to participate, or who do not wish to donate blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 antibodies in laboratory confirmed SARS-CoV-2 patients | Month 6
  To describe the immune response to SARS-CoV-2 infection by measuring the level of IgG and IgM in the blood of patients six months after laboratory-confirmed diagnosis of SARS-CoV-2
Seroprevalence of SARS-CoV-2 antibodies in laboratory confirmed SARS-CoV-2 patients | Month 12
  To describe the immune response to SARS-CoV-2 infection by measuring the level of IgG and IgM in the blood of patients 12 months after laboratory-confirmed diagnosis of SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Philippe VANHEMS, MD, Principal Investigator — Lyon, France, 69003
Locations (2):
- France (2):
  - Service épidémiologie, Hopital édouard Herriot, Lyon, Rhone
  - hopital Edouard Herriot, Lyon

REFERENCES:
- [Result] Khanafer N, Henaff L, Bennia S, Termoz A, Chapurlat R, Escuret V, Proriol M, Duvert F, Mena C, Planckaert C, Trehet-Mandez N, Saadatian-Elahi M, Vanhems P. Factors Associated with Long COVID-19 in a French Multicentric Prospective Cohort Study. Int J Environ Res Public Health. 2023 Aug 29;20(17):6678. doi: 10.3390/ijerph20176678. PMID 37681818